CLINICAL TRIAL: NCT00593853
Title: A Phase II, Randomized, Double-blind, Placebo Controlled Trial of Methylphenidate Hydrochloride for Reduction of Fatigue in Prostate Cancer Patients Receiving LHRH-Agonist Therapy
Brief Title: Efficacy Study of Methylphenidate Hydrochloride to Reduce Fatigue in Prostate Cancer Patients Receiving Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Dr. Neil Fleshner, MD, MPH, FRCSC, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEUPR_L_01; 07-0350-C
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Prostatic Neoplasms; Fatigue
Keywords: LHRH-agonist related fatigue
MeSH Terms: conditions — Prostatic Neoplasms; Fatigue | interventions — Methylphenidate; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Methylphenidate Hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Matched Placebo

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride — Run in period of 5mg QD,PO for 2 weeks followed by 5mg BID,PO for 8 weeks (full daily dose of 10mg). Followed by a 2 week taper period of 5mg QD,PO to complete 12 week cycle.
  Other Names: Ritalin
  Arms: 1
Drug: Matched Placebo — Run in period of 5mg QD,PO for 2 weeks followed by 5mg BID,PO for 8 weeks (full daily dose of 10mg). Followed by a 2 week taper period of 5mg QD,PO to complete 12 week cycle.
  Other Names: Inert Filler (lactose)
  Arms: 2

SUMMARY:
The purpose of this study is to determine if methylphenidate improves fatigue in men undergoing hormonal therapy for prostate cancer with an LHRH-agonist.

DETAILED DESCRIPTION:
This study will determine if methylphenidate improves fatigue in men undergoing hormonal therapy for prostate cancer. Fatigue is a common problem experienced by cancer patients. Those patients who are receiving chemotherapy or radiation are especially vulnerable to fatigue, as are men with prostate cancer who are receiving hormonal therapy with an LHRH-agonist (androgen deprivation therapy). Eligible men will be randomized to a daily dose of 10 mg methylphenidate or placebo for a total treatment period of 12 weeks. Subjects will be monitored for changes in fatigue and mood during this period. While the exact cause of fatigue in this setting is unknown, this study will hopefully lead to a better understanding of the process and provide patients with a much-needed remedy for fatigue

ELIGIBILITY:
Inclusion:

* Age > 18 and ≤ 85 years
* Histologically confirmed prostate cancer
* Currently receiving LHRH-agonist therapy for greater than 6 months with measurable fatigue, defined as a score of >1 on the Bruera global fatigue severity scale OR
* Deemed eligible to commence LHRH-agonist therapy, with confirmation of fatigue at Screening Visit 2
* Have a serum PSA which is stable or decreasing based on the PSA trend over the last 2 values taken at least 2 months apart, with the more recent value taken at least 2 months after initiation of LHRH-agonist therapy.
* Have adequate liver and renal function (Bilirubin ≤ 1.5 x ULN and AST, ALT and Serum Creatinine < 2 x ULN)
* Able to swallow and retain oral medication
* Life expectancy of at least 1 year
* Able to read and write in English (and therefore accurately complete the required study questionnaires), understand instructions related to study procedures and give written informed consent.

Exclusion:

* Current malignancy or received treatment for a previous malignancy within the last 3 years other than prostate cancer (other exceptions are superficial bladder cancer or non-melanoma skin cancer)
* Previous chemotherapy within the last 5 years
* Anemia (Hemoglobin < 100 g/L)
* Myocardial infarction within past 6 months
* Any unstable serious co-existing medical condition(s) including but not limited to ; unstable or poorly controlled coronary artery disease, chronic atrial fibrillation, uncontrolled hypertension, uncontrolled diabetes, Severe bleeding diseases or immune disorders
* Severe depression as defined by CES-D score >27
* History of motor tics, seizures or a family history of Tourette's syndrome
* Infection with HIV (Human Immunodeficiency Virus), HBV (Hepatitis B) or HCV (Hepatitis C)
* Evidence of drug or alcohol abuse
* Known hypersensitivity to methylphenidate
* Possess any other contraindications to methylphenidate use

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To assess the ability of methylphenidate 5 mg BID (10 mg daily) to reduce LHRH-agonist-related fatigue in prostate cancer patients as measured by the Functional Assessment of Cancer Therapy Fatigue subscale (FACT-F). | 3 months pre-treatment (LHRH-agnost naive group only), randomization, 6 weeks, 10 weeks, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Reduction in LHRH-agonist-related fatigue in prostate cancer patients as measured by the Bruera Global Fatigue Severity Scale | Screening Visit 1, 3 months pre-treatment (LHRH-agonist naive group only), Screening Visit 2 (LHRH-agonist naive group only), Randomization, 2 weeks, 6 weeks, 10 weeks, 12 weeks, 24 weeks
Reduction in LHRH-agonist-related fatigue in prostate cancer patients as measured by the Centre for Epidemiological Studies Depression Scale(CESD) | Screening Visit 1, 3 months pre-treatment (LHRH-agonist naive group only), Screening Visit 2 (LHRH-agonist naive group only), Randomization, 6 weeks, 10 weeks, 24 weeks
Reduction in LHRH-agonist-related fatigue in prostate cancer patients as measured by the Medical Outcomes Study 36-Item Short Form (SF-36) | 3 months pre-treatment (LHRH-agonist naive group only), Randomization, 6 weeks, 10 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil E Fleshner, MD, Principal Investigator — University Health Network, Toronto; Shabbir MH Alibhai, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- UHN Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Richard PO, Fleshner NE, Bhatt JR, Hersey KM, Chahin R, Alibhai SM. Phase II, randomised, double-blind, placebo-controlled trial of methylphenidate for reduction of fatigue levels in patients with prostate cancer receiving LHRH-agonist therapy. BJU Int. 2015 Nov;116(5):744-52. doi: 10.1111/bju.12755. Epub 2015 Jun 8. PMID 24684534